CLINICAL TRIAL: NCT04265534
Title: A Phase 2 Randomized, Multicenter, Double-Blind Study of the Glutaminase Inhibitor Telaglenastat With Pembrolizumab and Chemotherapy Versus Placebo With Pembrolizumab and Chemotherapy in First-Line, Metastatic KEAP1/NRF2-Mutated, Nonsquamous, Non-Small Cell Lung Cancer (NSCLC)
Brief Title: KEAPSAKE: A Study of Telaglenastat (CB-839) With Standard-of-Care Chemoimmunotherapy in 1L KEAP1/NRF2-Mutated, Nonsquamous NSCLC
Acronym: KEAPSAKE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Clinical Benefit
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX-839-014
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-Small Cell Lung Cancer; Non-squamous Non-small-cell Lung Cancer; Non-Squamous Non-Small Cell Neoplasm of Lung; KEAP1 Gene Mutation; NRF2 Gene Mutation; NFE2L2 Gene Mutation
Keywords: NSCLC; KEAP1; NRF2; NFE2l2; LKB1; STK11; Next Generation Sequencing; NGS; Mutation; Pembrolizumab; Pemetrexed; Carboplatin; Randomized; Placebo; Chemotherapy; Targeted Therapy; Telaglenastat; Glutamine; Glutaminase; Glutathione; Immunotherapy; Front-line; First-line; Non-squamous; Keytruda; Alimta; Guardant360
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — CB-839; Carboplatin; Pemetrexed; pembrolizumab; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telaglenastat with Pembrolizumab and Chemotherapy (Experimental): The glutaminase inhibitor telaglenastat will be administered orally, twice daily with food, every day in combination with standard-of-care pembrolizumab plus chemotherapy by intravenous (IV) infusion every 3 weeks.
  Interventions: Drug: Telaglenastat; Drug: Carboplatin Chemotherapy; Drug: Pemetrexed Chemotherapy; Biological: Pembrolizumab Immunotherapy; Dietary Supplement: Folic acid 400 -1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg
- Placebo with Pembrolizumab and Chemotherapy (Placebo Comparator): Placebo will be administered orally twice daily with food every day in combination with standard-of-care pembrolizumab plus chemotherapy by IV infusion every 3 weeks.
  Interventions: Drug: Carboplatin Chemotherapy; Drug: Pemetrexed Chemotherapy; Biological: Pembrolizumab Immunotherapy; Drug: Placebo; Dietary Supplement: Folic acid 400 -1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg

INTERVENTIONS:
Drug: Telaglenastat — Oral Glutaminase Inhibitor
  Other Names: CB-839
  Arms: Telaglenastat with Pembrolizumab and Chemotherapy
Drug: Carboplatin Chemotherapy — IV infusion
  Other Names: Paraplatin
Drug: Pemetrexed Chemotherapy — IV infusion
  Other Names: Alimta
Biological: Pembrolizumab Immunotherapy — IV infusion
  Other Names: Keytruda
Drug: Placebo — Oral placebo
  Other Names: Oral placebo
  Arms: Placebo with Pembrolizumab and Chemotherapy
Dietary Supplement: Folic acid 400 -1000 μg — Orally, once daily beginning 7 days prior to the first dose of pemetrexed and continue until 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 1000 μg — Vitamin B12 1000 μg Intramuscular injection one week prior to the first dose of pemetrexed and once every 3 cycles (9 weeks) thereafter. Subsequent vitamin B12 injections may be given the same day as pemetrexed administration.
Drug: Dexamethasone 4 mg — For prophylaxis, orally twice per day (or equivalent). Taken the day before, day of, and day after pemetrexed administration.

SUMMARY:
This is a Phase 2, randomized, multicenter, double-blind study of the glutaminase inhibitor telaglenastat with standard-of-care pembrolizumab and chemotherapy versus placebo with standard-of-care pembrolizumab and chemotherapy for first line treatment of metastatic disease in patients with KEAP1/NRF2-mutated, stage IV, nonsquamous, non-small cell lung cancer (NSCLC). The study primary endpoints are PFS per RECIST v. 1.1 and safety. KEAP1/NRF2 mutation status (for eligibility) and STK11/LKB1 status (for stratification) will be determined by next generation sequencing. A commercial liquid biopsy (circulating tumor DNA) NGS test will be provided to study participants free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented non-squamous NSCLC
2. Stage IV (M1a-c, AJCC 8th Edition, Amin 2017) disease not previously treated with systemic therapy for metastatic NSCLC

   a. Patients who received adjuvant or neo-adjuvant therapy (with or without immunotherapy) for localized NSCLC are eligible if all adjuvant/neo-adjuvant therapy (including immunotherapy) was completed at least 6 months prior to the development of metastatic disease.
3. No known actionable mutation in EGFR, ALK, ROS1, BRAF, NTRK or other known actionable mutation for which there is approved therapy in the first-line lung cancer setting
4. Must have at least one radiographically measurable lesion per RECIST v1.1 defined as a lesion that is ≥ 10 mm in longest diameter or lymph node that is ≥ 15 mm in short axis imaged by computed tomography (CT) scan or magnetic resonance imaging (MRI)

   a. Target lesions situated in a previously irradiated area may be considered measurable if progression has been demonstrated subsequent to radiation therapy
5. Age ≥ 18 years on the day of signing informed consent
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Estimated life expectancy of at least 3 months
8. Recovery to baseline or ≤ grade 1 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from toxicities related to the prior treatment, unless after discussion with the medical monitor, the AE(s) are deemed clinically non-significant and/or stable on supportive therapy
9. Has sponsor-approved eligible mutation in KEAP1 or NRF2 documented by NGS from a CAP-accredited and/or CLIA-certified laboratory (study-provided NGS or other NGS) and STK11 mutation status is known for the purpose of stratification.
10. Adequate organ function laboratory findings (defined per protocol)
11. Reproductive status:

    a. A female patient of childbearing potential must: i. Have a negative serum pregnancy test within 7 days prior to randomization ii. Agree to use methods of contraception outlined in Section 8.1.2 during the study through 120 days following the last dose of telaglenastat or pembrolizumab, or through 180 days following the last dose of chemotherapeutic drugs iii. Postmenopausal females (no menses for > 1 year without an alternate medical cause) and surgically sterilized females are exempt from these requirements b. Male patients who are sexually active with heterosexual partners of childbearing potential must agree to contraceptive requirements outlined in Section 8.1.2 and refrain from donating sperm during the study through 120 days following the last dose of telaglenastat or pembrolizumab, or through 180 days following the last dose of chemotherapeutic drugs

Exclusion Criteria:

1. Squamous cell histology and mixed histology tumors with any small-cell/neuroendocrine component (other mixed histology should be reviewed with the medical monitor for eligibility)
2. Any other concurrent malignancy requiring local or systemic therapy. Patients with other previously treated malignancy(ies) are allowed if the specific neoplasm, in the opinion of the principal investigator and with the agreement of the medical monitor, is not expected to interfere with study-specific endpoints
3. Radiation therapy to the lung > 30 Gy within 6 months prior to randomization
4. Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, abdominal carcinomatosis
5. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)

   a. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Treatment with chronic systemic steroids greater than 10 mg equivalent of prednisone per day
7. Unstable/inadequate cardiac function, defined as the following:

   1. Myocardial infarction or symptomatic ischemia within 6 months prior to randomization
   2. Uncontrolled or clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] are eligible)
   3. Congestive heart failure (New York Heart Association class III to IV)
8. Unable to swallow oral medications
9. Known sensitivity to any component of the study treatment (pembrolizumab, carboplatin, pemetrexed, and/or telaglenastat) or previous severe hypersensitivity to another monoclonal antibody (mAb)
10. Unable or unwilling to take folic acid or vitamin B12 supplementation (per pemetrexed label)
11. Unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) as specified in pemetrexed label
12. Interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoid treatment
13. Unable or unwilling to discontinue proton pump inhibitor (PPI) use ≥ 5 days prior to randomization
14. Patient known to be positive for Human Immunodeficiency Virus (HIV)
15. Known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hepatitis C antibody result and known quantitative Hepatitis C virus RNA results greater than the lower limits of detection of the assay. Patients receiving antiviral therapy for Hepatitis B or C also are not eligible
16. Any condition including social, psychiatric or medical (including uncontrolled significant concurrent illness) that in the opinion of the Investigator could interfere with treatment or protocol-related procedures
17. Regular use of illicit drugs or history (within past year) of substance abuse (including alcohol)
18. Patients who are pregnant or lactating
19. Major surgery < 3 weeks prior to randomization. In addition, patients with ongoing clinically relevant complications from prior surgery are not eligible and they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
20. Any radiation therapy within 2 weeks prior to randomization (with exception of SRS for brain metastases). In addition, patients with ongoing clinically relevant complications from prior radiation therapy, patients requiring corticosteroids to treat radiation toxicity and patients who developed radiation pneumonitis are not eligible.
21. Symptomatic ascites or pleural effusion. Patients who are clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) are eligible
22. Refractory nausea and vomiting, uncontrolled diarrhea, malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes or other situation that may preclude adequate absorption or oral study drug
23. Infection requiring more than 5 days of parenteral antibiotics, antivirals, or antifungals within two weeks prior to randomization. Anti-infective therapy must be completed at least 7 days before randomization
24. Patients with active and/or untreated central nervous system metastasis including carcinomatous meningitis (leptomeningeal disease) are not eligible. Patients with previously treated brain metastases are eligible if they meet the following criteria:

    1. Received definitive treatment with stereotactic radiosurgery (SRS) or surgery to all known central nervous system (CNS) lesions (whole brain radiotherapy is not an eligible modality)
    2. Be at least 4 weeks post-surgical resection of CNS disease, symptomatically stable and off steroids before randomization
25. Any live-virus vaccination within 28 days prior to randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist ®) are live attenuated vaccines and are not allowed
26. Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS), Assessed by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 24 months
  Duration of investigator-determined PFS per RECIST v1.1 in the intent-to-treat (ITT) population
Safety and Tolerability of Telaglenastat Plus Standard-of-Care Pembrolizumab and Chemotherapy Assessed by Type, Incidence, Severity, Seriousness, and Study Drug Relatedness of Adverse Events per CTCAE v5.0 | Up to 55 months
Recommended Phase 2 Dose of Telaglenastat in Combination with Standard-of-Care Pembrolizumab and Chemotherapy Assessed by Incidence and Nature of Protocol Defined Dose-Limiting Toxicities (DLTs) During the Safety Run-in Period | Up to 6 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) for Patients Treated with Telaglenastat plus Standard-of-Care Pembrolizumab and Chemotherapy versus Placebo plus Standard-of-Care Pembrolizumab and Chemotherapy | Up to 24 months
  ORR is defined as the percentage of patients with complete response (CR) or partial response (PR) according to the RECIST v1.1 criteria as assessed by the investigator.
Duration of Response (DOR) for Patients Treated with Telaglenastat plus Standard-of-Care Pembrolizumab and Chemotherapy versus Placebo plus Standard-of-Care Pembrolizumab and Chemotherapy | Up to 24 months
  DOR is defined as the duration of response for patients achieving a CR or PR
Overall Survival | Up to 55 months
PFS in the Subgroup of Patients with Biochemical Evidence of Activation of the NRF2 Pathway | Up to 24 months
ORR in the Subgroup of Patients with Biochemical Evidence of Activation of the NRF2 Pathway | Up to 24 months
DOR in the Subgroup of Patients with Biochemical Evidence of Activation of the NRF2 Pathway | Up to 24 months
OS in the Subgroup of Patients with Biochemical Evidence of Activation of the NRF2 Pathway | Up to 55 months

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kuriakose, MD, Study Director — Calithera Biosciences, Inc
Locations (102):
- United States (102):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama - Mitchell Cancer Center, Mobile, Alabama
  - Yuma Regional Medical Center, Yuma, Arizona
  - Compassionate Cancer Care, Fountain Valley, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of California Irvine, Chao Family Comprehensive Cancer Center, Orange, California
  - St. Joseph Heritage Healthcare - Santa Rosa, Santa Rosa, California
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital Lynn Cancer Institute, Boca Raton, Florida
  - Holy Cross Hospital - Bines Cancer Center, Fort Lauderdale, Florida
  - Florida Cancer Specialist - South (SCRI), Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Hollywood, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Cancer Specialist - North (SCRI), St. Petersburg, Florida
  - Florida Cancer Specialist - Panhandle (SCRI), Tallahassee, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialist - East (SCRI), West Palm Beach, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwest Georgia Oncology, Marietta, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Oncology of Northshore, Rolling Meadows, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Beacon Health, South Bend, Indiana
  - University of Kansas Medical Center (KUMC), Westwood, Kansas
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Johns Hopkins Bayview Memorial Hospital, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology - USOR, Columbia, Maryland
  - Frederick Health - James M. Stockman Cancer Institute, Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Bronson Methodist Hospital (West Michigan Cancer Center), Kalamazoo, Michigan
  - St. Joseph Mercy Hospital Cancer Care Center, Ypsilanti, Michigan
  - Minnesota Oncology Hematology, P.A., Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Oncology Hematology, P.A., Saint Paul, Minnesota
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Washington University, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New Jersey Cancer Care and Blood Disorders (NJCCBD), Belleville, New Jersey
  - Summit Medical Group, Berkeley Heights, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. (400 Patoon Creek Blvd.), Albany, New York
  - New York Oncology Hematology, P.C. (43 New Scotland Ave.), Albany, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - Pelmutter Cancer Center at Winthrop, Mineola, New York
  - New York University Langone (NYU), New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Cone Health at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Aultman Hospital, Canton, Ohio
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Ohio State University, James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Ohio Health, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Oklahoma Cancer Specialists and Research Institute (OCSRI), Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health & Science University (OHSU) Knight Cancer Institute, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Pennsylvania State University Milton S. Hershey Medical Center, State College, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Tennessee Oncology - Chattanooga (SCRI), Chattanooga, Tennessee
  - Tennessee Oncology - Nashville (SCRI), Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology Beaumont - USOR, Beaumont, Texas
  - Texas Oncology - Denison, Denison, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Oncology Consultants, Houston, Texas
  - Oncology and Hematology of South Texas, Laredo, Texas
  - Utah Cancer Specialist, Salt Lake City, Utah
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Oncology and Hematology Associates of Southwest Virginia, Blacksburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Low Moor, Virginia
  - Virginia Commonwealth University (VCU) Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Salem, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Wytheville, Virginia
  - University of Washington Seattle Cancer Care Alliance (SCCA), Seattle, Washington
  - Northwest Medical Specialities, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin (MCW), Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179